CLINICAL TRIAL: NCT03304288
Title: The Combination of Low-dose Rituximab and All-trans Retinoic Acid as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia: a Multicenter, Randomized, Open-label Trial
Brief Title: The Combination of Low-dose Rituximab and ATRA as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Navy General Hospital, Beijing (Other); Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Xiao-hui Zhang, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81670116
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Immune Thrombocytopenia
Keywords: all-trans retinoid acid; rituximab; steroid-resistant; refractory; low-dose
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; Tretinoin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low-dose rituximab & ATRA (Experimental): rituximab 100mg once weekly for 6 weeks and oral all-trance retinoid acid 20mg/m^2 qd for 12 weeks.
  Interventions: Drug: Rituximab; Drug: All-trans retinoic acid
- low-dose rituximab (Active Comparator): rituximab 100mg once weekly for 6 weeks
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Low-dose rituximab was used in combination with ATRA or as the monotherapy
Drug: All-trans retinoic acid — ATRA was used in combination with low-dose rituximab
  Arms: low-dose rituximab & ATRA

SUMMARY:
Randomized, open-label, multicentre study to assess the efficacy and safety of the combination of low-dose rituximab and ATRA in patients with steroid-resistant/relapsed ITP.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a severe bleeding disorder. Approximately 2/3 of patients achieve remission from first-line therapies. However, the underlying mechanism of steroid-resistant or relapsed ITP is not well understood; thus, treatment remains a great challenge. Rituximab has been shown to partly improve the complete remission rate of ITP. All-trans retinoic acid (ATRA) has an immunomodulatory effect on haematopoiesis, making it a possible treatment option.

A multicentre prospective study was performed in non-splenectomized ITP patients who were either resistant to a standard dose of corticosteroids or had relapsed. Patients were randomized to the low-dose rituximab+ATRA and the low-dose rituximab monotherapy groups. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Interim analysis was scheduled at 50% through recruitment. Adverse events are also recorded throughout the study, in order to assess the efficacy and safety of the combination of low-dose rituximab and ATRA in patients with steroid-resistant/relapsed ITP.

ELIGIBILITY:
Inclusion Criteria:

* ITP confirmed by excluding other supervened causes of thrombocytopenia;
* Platelet count of less than 30×10^9/L at enrollment;
* Patients who did not achieve a sustained response to treatment with full dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation;
* ECOG<2.

Exclusion Criteria:

* Secondary immune thrombocytopenia (e.g., patients with HIV, HCV, Helicobacter pylori infection or patients with systemic lupus erythematosus)
* Congestive heart failure
* Severe arrhythmia
* Nursing or pregnant women
* Aspartate aminotransferase and alanine transaminase levels ≥ 3×the upper limit of the normal threshold criteria
* Creatinine or serum bilirubin levels each 1•5 times or more than the normal range
* Active or previous malignancy
* Patients with other diseases were undergoing treatment with immunosuppressants
* Patients with ITP had received rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
overall response | From the start of study treatment (Day 1) up to the end of Year 1
  The number of participants (responders) with platelet count >=30x10^9/L and at least a 2-fold increase in the baseline count (PR) or a platelet count >=100x10^9/L (CR) and the absence of bleeding, without rescue medication at 1-year follow-up. Interim analysis was scheduled at 50% through recruitment.
sustained response | From the start of study treatment (Day 1) up to the end of Year 1
  The number of participants that can maintain the platelet count > 30 x 109/L, an absence of bleeding events, and without requirement for any other ITP-specific treatment for 6 consecutive months after achievement of response. Interim analysis was scheduled at 50% through recruitment.

SECONDARY OUTCOMES:
complete response | From the start of study treatment (Day 1) up to the end of Year 1
  The number of participants (responders) with platelet count>=100x10^9/L (CR) and the absence of bleeding, without rescue medication at 1-year follow-up. Interim analysis was scheduled at 50% through recruitment.
time to response | From the start of study treatment (Day 1) up to the end of Year 1
  Time to response was defined as the time from starting treatment to the time to achieve the response. Interim analysis was scheduled at 50% through recruitment.
duration of response | From the start of study treatment (Day 1) up to the end of Year 1
  Duration of response was measured from the achievement of response to the loss of response. Interim analysis was scheduled at 50% through recruitment.
incidence of adverse events | From the start of study treatment (Day 1) up to the end of Year 1
  All patients were assessed for adverse events every week during the first 4 weeks of treatment, and at 2-weeks interval for the following 5 months, and monthly thereafter. Adverse events were scaled according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Interim analysis was scheduled at 50% through recruitment.
Initial response | From the start of study treatment (Day 1) up to the end of Week 4
  The number of patients who achieve response at 4 weeks following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-hui Zhang, Professor, Principal Investigator — Peking University Insititute of Hematology, Peking University People's Hospital
Locations (4):
- China (4):
  - Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality
  - Navy General Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Wu YJ, Liu H, Zeng QZ, Liu Y, Wang JW, Wang WS, Jia-Feng, Zhou HB, Huang QS, He Y, Fu HX, Zhu XL, Jiang Q, Jiang H, Chang YJ, Xu LP, Huang XJ, Zhang XH. All-trans retinoic acid plus low-dose rituximab vs low-dose rituximab in corticosteroid-resistant or relapsed ITP. Blood. 2022 Jan 20;139(3):333-342. doi: 10.1182/blood.2021013393. PMID 34665865